CLINICAL TRIAL: NCT04209400
Title: A Comparative Randomized Double-Blind Study of Safety and Immunogenicity of Recombinant Hepatitis B Vaccine Sci-B-Vac® in Adult Study Subjects
Brief Title: Safety and Immunogenicity of Recombinant Hepatitis B Vaccine Sci-B-Vac® Compared to Engerix-B®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 38-13-040 RUS
Record Dates: First submitted 2019-12-09; First posted 2019-12-24 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B
Keywords: Sci-B-Vac®; Prophylactic vaccine; HepB vaccines; Phase 3; pre-S1; pre-S2; Surface antigen
MeSH Terms: conditions — Hepatitis B | interventions — Pre-S vaccine; Engerix-B

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sci-B-Vac® (Experimental): The 3-antigen HepB vaccine, Sci-B-Vac® contains three recombinant proteins of HBV viral envelope: small S, medium pre-S2, and large pre-S1 surface antigens. Sci-B-Vac® was supplied in 1.0 ml vials.
  Interventions: Biological: Sci-B-Vac®
- Engerix-B® (Active Comparator): The single-antigen HepB vaccine, Engerix-B® (GSK), contains the small S recombinant protein. Engerix-B® was supplied in 1.0 ml vials.
  Interventions: Biological: Engerix-B®

INTERVENTIONS:
Biological: Sci-B-Vac® — Sci-B-Vac® vaccine-10 μg of HBsAg, intramuscular injection of 10 μg/ml
  Arms: Sci-B-Vac®
Biological: Engerix-B® — Engerix-B® vaccine-20 μg of HBsAg, intramuscular injection of 20 μg/ml
  Arms: Engerix-B®

SUMMARY:
This study was a comparative, randomized, double-blind clinical study of the efficacy and safety of Sci-B-Vac® (10 μg dose) and the Engerix-B® (20 μg dose) vaccines in two parallel groups of hepatitis B-naive healthy adult subjects in Russia.

DETAILED DESCRIPTION:
This study was a comparative randomized double-blind clinical study of the efficacy and safety of Sci-B-Vac® (10 μg dose) and the Engerix-B® (20 μg dose) vaccines in hepatitis B-naive healthy adult subjects (n = 100). The study was conducted at 3 study sites in the Russian Federation. Subjects who passed the screening successfully were randomized into two groups, Sci-B-Vac® (10 μg dose) and Engerix-B® (20 μg dose), in a 1:1 ratio. Subjects were vaccinated three times at days 1, 28, and 180 of the study.

Statistical Methods: Evaluation and comparison of immunogenicity were conducted at baseline, day 28, day 90 (60 days after the second vaccination), day 180 (prior to administering the third vaccine, 90 days after the second vaccination), and day 210 (30 days after the third vaccination) of the study.

The primary outcome was the seroconversion rate (proportion of subjects with anti-HBs levels ≥ 2.1 mIU/mL) after the third vaccination at day 210. The non-inferiority margin was set at 4%. The percentage of subjects who achieved seroconversion was analyzed using the Chi-square test for proportions along with the McNemar's test for repeated measurements in each group. The non-inferiority hypotheses were confirmed if the lower range of the confidence interval was at least -4%. The secondary endpoint was SPR (≥10 mIU/ml), measured at days 1, 28, 90, 180 and 210.

Demographic data, initial parameters, safety parameters, tolerance of the experimental vaccine, and other study parameters were analyzed using descriptive statistics (mean value, standard deviation, median, minimum and maximum values, range, quartiles, the number of valid cases-for quantitative variables; absolute number, proportion, allocation-for qualitative variables). A comparative assessment of the detection rate for different parameters in the two comparison groups was conducted using the Student's t-test; differences were considered statistically significant at a significance level of 5%. The assay used to measure anti-HBs concentrations had an upper limit of 1000 mIU/mL.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written Informed Consent to participate in the study from the subject.
2. Male or female between 18 and 45 years old without previous contact with hepatitis B virus (HBV).
3. Good health condition based on full physical examination.
4. Normal values of laboratory biochemical blood tests.
5. Seronegative with respect to anti-HBs (surface) antibodies, anti-HBc (core) antibodies, and HBs Antigen (HBsAg) on screening.
6. Not pregnant and not breast-feeding.
7. For men and women of reproductive age: consent for use of an effective contraception method, for example, an intrauterine device, oral contraceptive, hypodermic implant or double barrier method (a condom with contraceptive sponge or contraceptive suppository) throughout the entire study.

Exclusion Criteria:

1. Congenital or inherited immunodeficiency disorder in family history.
2. Information of a serious blood disorder, cardiac disorder, or tumour.
3. Current use of any medication that could alter immune reactivity.
4. Infection with HBV at the present time or in the past, confirmed by HBV markers test.
5. Anaphylaxis or severe allergy, or atopy, history of alcoholism or drug abuse.
6. Pregnancy and breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04-18 (Actual); Primary Completion 2015-04-20 (Actual); Study Completion 2015-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Esaulenko, Principal Investigator — Saint Petersburg State Paediatric Medical University
Locations (1):
- Saint Petersburg State Budgetary Healthcare Institution, Saint Petersburg, Mirgorodskaya, Russia

REFERENCES:
- [Result] Esaulenko EV, Yakovlev AA, Volkov GA, Sukhoruk AA, Surkov KG, Kruglyakov PV, Diaz-Mitoma F. Efficacy and Safety of a 3-Antigen (Pre-S1/Pre-S2/S) Hepatitis B Vaccine: Results of a Phase 3 Randomized Clinical Trial in the Russian Federation. Clin Infect Dis. 2021 Nov 2;73(9):e3333-e3339. doi: 10.1093/cid/ciaa1649. PMID 33119068

RESULTS

PARTICIPANT FLOW:
Groups:
- Sci-B-Vac®: Sci-B-Vac® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 10ug, IM injection at Days 1, 28 and 180 Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
- Engerix-B®: Engerix-B® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 20ug, IM injection at Days 0, 28, and 180.
  Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
Period: Overall Study
Arm/Group | Sci-B-Vac® | Engerix-B®
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sci-B-Vac®: Sci-B-Vac® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 10ug, IM injection at Days 0, 28, and 180.
  Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
- Total: Total of all reporting groups
Arm/Group | Sci-B-Vac® | Engerix-B® | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.38 (7.72) | 30.56 (8.13) | 29.47 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 18 | 21 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian-Russians | 50 | 50 | 100
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate
Description: Percentage of subjects with an anti-HBs antibody level ≥ 2.1 mIU/mL 30 days after the last of three vaccinations. Seroconversion is defined as the development of a detectable anti-HBs antibody level above an established threshold of 2.1 mIU/mL.
Time Frame: Day 210
Population: The primary analysis was performed on the intent-to-treat (ITT) set, which included all participants randomized. Analysis of the study parameters for vaccine immunogenicity was performed for all subjects included in the vaccine groups who received at least one injection, if at least one assessment after the start of the vaccination was available.
Measure: Count of Participants; unit: Participants
Groups:
- Sci-B-Vac®: Sci-B-Vac® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 10ug, intramuscular (IM) injection at Days 0, 28, and 180.
  Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
- Engerix-B®: Engerix-B® (hepatitis B vaccine) Hepatitis B Vaccination, Solution, 20ug, intramuscular (IM) injection at Days 0, 28, and 180.
  Hepatitis B Vaccination: Prophylactic Hepatitis B Vaccination
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 47 | 47
Participants | 47 | 46
Statistical Analysis 1: Comparison: Sci-B-Vac® vs Engerix-B®; The null hypothesis is that the vaccines equally affect the achievement of seroconversion level; Test type: Non-Inferiority — P < 0.05 is considered a statistically significant difference in seroconversion between the two groups; p = 1, Chi-squared

2. Secondary Outcome: Seroprotection Rate
Description: Percentage of subjects with an anti-HBs antibody level ≥ 10 mIU/mL prior to vaccination, 28 days after the first vaccination, 60 and 150 days after the second vaccination and 30 days after the third vaccination. The development of an anti-HBs antibody level of at least 10 mIU/mL is an established surrogate of seroprotection and correlate of protective immunity against HBV.
Time Frame: Days 1, 28, 90, 180, 210
Population: The analysis was performed on the intent-to-treat (ITT) set, which included all participants randomized. Analysis of the study parameters for vaccine immunogenicity was performed for all subjects included in the vaccine groups who received at least one injection, if at least one assessment after the start of the vaccination was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
Participants
  Day 1 | 0 | 0
  Day 28: number analyzed (Participants) | 49 | 47
  Day 28 | 30 | 24
  Day 90: number analyzed (Participants) | 49 | 47
  Day 90 | 47 | 41
  Day 180: number analyzed (Participants) | 47 | 47
  Day 180 | 47 | 42

3. Secondary Outcome: Seroconversion Rate
Description: Percentage of subjects with an anti-HBs antibody level ≥ 2.1 mIU/mL prior to vaccination, 28 days after the first vaccination and 60 and 150 days after the second vaccination. Seroconversion is defined as the development of a detectable anti-HBs antibody level above an established threshold of 2.1 mIU/mL.
Time Frame: Days 1, 28, 90, 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
Participants
  Day 1 | 0 | 0
  Day 28: number analyzed (Participants) | 49 | 47
  Day 28 | 46 | 36
  Day 90: number analyzed (Participants) | 48 | 47
  Day 90 | 48 | 45
  Day 180: number analyzed (Participants) | 47 | 47
  Day 180 | 47 | 45

4. Secondary Outcome: Geometric Mean Concentrations (GMC) of HBs Antibodies
Description: Geometric mean concentration of anti-HBs antibody in mIU/mL 28 days after the first vaccination, 60 and 150 days after the second vaccination, and 30 days after the third vaccination.
Time Frame: Days 1, 28, 90, 180, and 210
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
mIU/mL
  Day 90 | 618.3 (404.2) | 378.7 (417.9)
  Day 180 | 757.7 (378.0) | 441.3 (437.6)
  Day 210 | 891.4 (253.7) | 787.0 (351.9)

5. Other Pre Specified Outcome: Adverse Events: Local Reactions at the Injection Site- Incidence of Redness
Description: Incidence of mild erythema at the injection site 1, 2 and 28 days after the first vaccination.
Time Frame: Day 1, Day 2, and Day 28
Population: The analysis of safety and tolerability was conducted in the population of subjects included in the study meeting the inclusion criteria while complying with the exclusion criteria, who received at least one dose of the experimental vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
Participants
  Day 1 | 8 | 4
  Day 2 | 2 | 1
  Day 28 | 3 | 0

6. Other Pre Specified Outcome: Adverse Events: Local Reactions at the Injection Site - Incidence of Itch
Description: Incidence of itchiness at the injection site at any point throughout the trial. Itchiness was assessed for 5 days following vaccinations on Days 1, 28, and 180 and also assessed on Day 90 and Day 210.
Time Frame: Days 1-5, Days 28-32, Day 90, Days 180-185, Day 210
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
Participants | 1 | 0

7. Other Pre Specified Outcome: Adverse Events: Local Reactions at the Injection Site - Incidence of Pain
Description: Incidence of pain at the injection site on the day of vaccination. Vaccination was performed on Day 1, Day 28, and Day 180.
Time Frame: Days 1, 28, 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
Participants
  Day 1 | 7 | 8
  Day 28 | 8 | 7
  Day 180 | 7 | 11

8. Other Pre Specified Outcome: Adverse Events: Local Reactions at the Injection Site - Intensity of Pain
Description: Pain was evaluated 30 minutes after each vaccination by the subject using the visual analogue scale. A higher score indicates greater pain intensity.
Time Frame: Days 1, 28, 180
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac® | Engerix-B®
Number analyzed (Participants) | 50 | 49
Participants
  Day 1 : Pains score 1 | 43 | 41
  Day 1 : Pain score 2 | 5 | 6
  Day 1 : Pain score 3 | 2 | 2
  Day 28 : Pain score 1: number analyzed (Participants) | 50 | 48
  Day 28 : Pain score 1 | 42 | 41
  Day 28 : Pain score 2: number analyzed (Participants) | 50 | 48
  Day 28 : Pain score 2 | 7 | 6
  Day 28 : Pain score 3: number analyzed (Participants) | 50 | 48
  Day 28 : Pain score 3 | 1 | 1
  Day 180 : Pain score 1: number analyzed (Participants) | 47 | 47
  Day 180 : Pain score 1 | 40 | 36
  Day 180 : Pain score 2: number analyzed (Participants) | 47 | 47
  Day 180 : Pain score 2 | 7 | 9
  Day 180 : Pain score 3: number analyzed (Participants) | 47 | 47
  Day 180 : Pain score 3 | 0 | 2

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 7 months.
Description: An AE is any unfavourable sign (including abnormal lab results), symptom, or disease that are time-associated with vaccine use, regardless whether or not they are viewed as having been caused by medicinal products, and whether they are mild or serious. Intensity of the adverse events were defined as Mild: Adverse event that is easily tolerated. Moderate: AEs causing discomfort sufficient for impairment of everyday activity. Severe: Adverse event preventing normal everyday activity
Arm/Group | Sci-B-Vac® | Engerix-B®
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 2/50 | 7/49
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sci-B-Vac® (N=50) | Engerix-B® (N=49)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
drowsiness (Nervous system disorders) | 2 (3) | 2 (2)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
metallic taste (Nervous system disorders) | 0 (0) | 1 (2)
acute respiratory viral infection (Infections and infestations) | 0 (0) | 1 (3)
rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Final CSR does not follow ICH guidelines and the original document in Russian was translated into English for the purpose of writing the manuscript and completing the documentation in clinicaltrials.gov

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No